CLINICAL TRIAL: NCT00147225
Title: Phase I/II Study of AMG 531 in Patients With Advanced Malignancy Receiving Treatment With Carboplatin
Brief Title: AMG 531 in Patients With Advanced Malignancy Receiving Treatment With Carboplatin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2005-0099
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Solid Tumors; Advanced Cancer
Keywords: Advanced Cancer; Advanced Malignancy; Solid Tumors; Thrombocytopenia; AMG 531; Romiplostim; Carboplatin; Paraplatin; Platelets; Adriamycin; Doxorubicin; Rubex; Ifosfamide; Ifex
MeSH Terms: conditions — Thrombocytopenia | interventions — romiplostim; Carboplatin; Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 mcg/kg AMG 531 Post Chemotherapy (Experimental): Cycle 1, Chemotherapy alone (Control Cycle); Beginning Cycle 2, Chemotherapy followed by 1 mcg/kg AMG 531 subcutaneously on day after chemotherapy and 2 days later (study cycle) of 21-28 day treatment cycle.
  Chemotherapy :
  1. Carboplatin [area under the concentration curve (AUC) = 11]; or
  2. Adriamycin - Ifosfamide (AI) regimen [Adriamycin 75-90 mg/m^2 intravenous (IV), Ifosfamide 10-14 gm/m^2 IV]; or
  3. High dose Ifosfamide: 14 gm/m^2.
  Interventions: Drug: AMG 531; Drug: Carboplatin; Drug: Adriamycin; Drug: Ifosfamide
- 3 mcg/kg AMG 531 Post Chemotherapy (Experimental): Cycle 1, Chemotherapy alone (Control Cycle); Beginning Cycle 2, Chemotherapy followed by 3 mcg/kg AMG 531 subcutaneously on day after chemotherapy and 2 days later (study cycle) of 21-28 day treatment cycle.
  Chemotherapy :
  1. Carboplatin [area under the concentration curve (AUC) = 11]; or
  2. AI regimen [Adriamycin 75-90 mg/m^2 intravenous (IV), Ifosfamide 10-14 gm/m^2 IV]; or
  3. High dose Ifosfamide: 14 gm/m^2.
  Interventions: Drug: AMG 531; Drug: Carboplatin; Drug: Adriamycin; Drug: Ifosfamide
- 10 mcg/kg AMG 531 Post Chemotherapy (Experimental): Cycle 1, Chemotherapy alone (Control Cycle); Beginning Cycle 2, Chemotherapy followed by 10 mcg/kg AMG 531 subcutaneously on day after chemotherapy and 2 days later (study cycle) of 21-28 day treatment cycle.
  Chemotherapy :
  1. Carboplatin [area under the concentration curve (AUC) = 11]; or
  2. AI regimen [Adriamycin 75-90 mg/m^2 intravenous (IV), Ifosfamide 10-14 gm/m^2 IV]; or
  3. High dose Ifosfamide: 14 gm/m^2.
  Interventions: Drug: AMG 531; Drug: Carboplatin; Drug: Adriamycin; Drug: Ifosfamide
- 10 mcg/kg Pre/Post Chemotherapy (Experimental): Cycle 1, Chemotherapy (Control Cycle); Beginning Cycle 2, 10 mcg/kg AMG 531 subcutaneously on Day -5 (pre dose) and on day after chemotherapy (post dose) of 21-28 day treatment cycle.
  Chemotherapy :
  1. Carboplatin [area under the concentration curve (AUC) = 11]; or
  2. AI regimen [Adriamycin 75-90 mg/m^2 intravenous (IV), Ifosfamide 10-14 gm/m^2 IV]; or
  3. High dose Ifosfamide: 14 gm/m^2.
  Interventions: Drug: AMG 531; Drug: Carboplatin; Drug: Adriamycin; Drug: Ifosfamide
- 5 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy (Experimental): Cycle 1, Chemotherapy alone (Control Cycle); Beginning Cycle 2, Chemotherapy followed by 5 mcg/kg AMG 531 for 2 doses on Days -5 and -3 (pre doses) and on day after chemotherapy and 2 days later (post doses) of 21-28 day treatment cycle.
  Chemotherapy :
  1. Carboplatin [area under the concentration curve (AUC) = 11]; or
  2. AI regimen [Adriamycin 75-90 mg/m^2 intravenous (IV), Ifosfamide 10-14 gm/m^2 IV]; or
  3. High dose Ifosfamide: 14 gm/m^2.
  Interventions: Drug: AMG 531; Drug: Carboplatin; Drug: Adriamycin; Drug: Ifosfamide
- 10 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy (Experimental): 10 mcg/kg AMG 531 + Pre/Pre/Post/Post Chemotherapy Cycle 1, Chemotherapy alone (Control Cycle); Beginning Cycle 2, Chemotherapy followed by 10 mcg/kg AMG 531 for 2 doses on Days -5 and -3 (pre doses) and on day after chemotherapy and 2 days later (post doses) of 21-28 day treatment cycle.
  Chemotherapy :
  1. Carboplatin [area under the concentration curve (AUC) = 11]; or
  2. AI regimen [Adriamycin 75-90 mg/m^2 intravenous (IV), Ifosfamide 10-14 gm/m^2 IV]; or
  3. High dose Ifosfamide: 14 gm/m^2.
  Interventions: Drug: AMG 531; Drug: Carboplatin; Drug: Adriamycin; Drug: Ifosfamide

INTERVENTIONS:
Drug: AMG 531 — Beginning with Cycle 2, administered in one of two schedules, either on day after chemotherapy and 2 days later (study cycle) or on day -5 (pre dose) and on day after chemotherapy (post dose) or combination of pre/post days of 21-28 day treatment cycle. Combination if Optimal biological dose (OBD) not reached, additional treatment at 10 mcg/kg dose level, with AMG 531 administered on day -5 (pre dose) and on day after chemotherapy (post dose).
  1, 3, or 10 mcg/kg given as injection under the skin (subcutaneous)
  Other Names: Romiplostim
Drug: Carboplatin — AUC=11; Cycle 1 chemotherapy alone then 3 weeks later, in Cycle 2, same dose of chemotherapy followed by AMG 531.
  Other Names: Paraplatin
Drug: Adriamycin — 75-90 mg/m^2 IV
  Other Names: Doxorubicin; Rubex
Drug: Ifosfamide — 10 gm/m^2 IV; OR, High dose ifosfamide = 14 gm/m^2.
  Other Names: Ifex

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of AMG 531 that will decrease the risk and severity of thrombocytopenia (low platelet counts) in patients who have received chemotherapy. Researchers will also look at the safety and effectiveness of AMG 531 (Romiplostim).

Primary Objectives:

1. To determine the clinical safety and tolerability of AMG 531 administered following chemotherapy in patients with advanced malignancy
2. To determine an optimal biologic dose (OBD) of AMG 531 administered in patients receiving chemotherapy known to cause severe thrombocytopenia
3. To evaluate the effects of AMG 531 on the degree and duration of thrombocytopenia and platelet recovery following chemotherapy

Secondary Objective:

1. To evaluate limited pharmacokinetics of AMG 531 administered by S.C. route post-chemotherapy

DETAILED DESCRIPTION:
Platelets are cells that help make the blood clot. A decrease in platelets can cause bleeding, which may prevent or delay a patient from receiving chemotherapy. Researchers want to find out if AMG 531 can lower the risk and severity of this side effect. AMG 531 is a protein that stimulates platelet production.

If you are eligible to take part in this study, you will be assigned to 1 of 6 dosing schedules of study drug. The dose of AMG 531 that you receive will depend on when you are enrolled.

In Cycle 1, all patients will receive chemotherapy by itself. Three (3) weeks later, in Cycle 2, the same dose of chemotherapy will be given followed by AMG 531. AMG 531 will be given on one of 3 schedules. AMG 531 will be given as an injection under the skin on the day after chemotherapy and 2 days later; it will be given 5 days before and the day after chemotherapy; or it will be given 5 and 3 days before chemotherapy and on the day after chemotherapy and 2 days later. The schedule you receive will depend on when you enroll on the study. After 2 cycles of treatment, based on response of the disease and tolerance to the treatment, all participants may be able to receive up to 4 more cycles of chemotherapy followed by AMG 531. All participants will continue on the same schedule you were receiving before. The dose of AMG 531 may be increased at one time point during the study based on the response of the platelet counts.

The number of blood tests drawn (about 3 teaspoons each) will depend on your clinical condition. These samples will be taken at least 2 times a week and as often as once a day during portions of the study. You will also have blood (about 1 teaspoon) collected for the evaluation of anti-AMG 531 antibody status before treatment starts, at the end of Cycles 2 and 4, and at the end of study.

You will be taken off the study if your disease gets worse or intolerable side effects occur. At the end of the study, you will have a medical history and physical exam, including measurement of vital signs. You will also have blood (about 1 teaspoon) drawn for routine tests.

This is an investigational study. AMG 531 is not FDA approved or commercially available. At this time, it is being used for research purposes only. Up to 56 patients will take part in this study. All will be enrolled at University of Texas (UT)MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of solid tumors who are at high risk for chemotherapy-induced severe thrombocytopenia related to the following regimens: (a) Carboplatin (AUC=11); (b) AI regimen (adriamycin 75-90mg/m2, Ifosfamide 10gm/m2); (c) High dose Ifosfamide (14gm/m2)
2. Age >/= 18 years.
3. Adequate hematologic (Absolute neutrophil count (ANC) >/= 1500/mm^3, platelet count >/= 100 x 10^9/L and Hgb >/= 8 gm/dL), renal (serum creatinine </= 2.0 mg/dL), and hepatic functions (total bilirubin </= 2 times, aspartate aminotransferase (AST or SGOT) or alanine aminotransferase (ALT or SGPT) </= 3 times the upper limit of the respective normal range).
4. Karnofsky Performance Status >/= 80
5. Signed informed consent form
6. Patients with childbearing potential (defined as not post-menopausal for 12 months or no previous surgical sterilization) must have a negative pregnancy test and use adequate birth control. [i.e. oral contraceptives, spermicide with either a condom, diaphragm or cervical cap, use of an intrauterine device (IUD), or abstinence].

Exclusion Criteria:

1. Patients with rapidly progressive disease (such as patients with rapidly accumulating ascites or pleural effusion).
2. Patients with hematologic malignancies.
3. Pregnant or lactating women.
4. History of central nervous system (CNS) metastasis.
5. Patients with significant cardiac disease (New York Hearth Association (NYHA) Class III or IV), dysrrhythmia, or recent history of MI or ischemia, transient ischemic attack or cerebrovascular accident (CVA), within the previous 6 months of study entry.
6. Patients with a history of thromboembolic events (history of deep venous thrombosis (DVT) or pulmonary embolus).
7. Prior chemotherapy, immunotherapy, or experimental drug (not FDA-approved drug) within 3 weeks. Patients will be eligible if day 1 of chemotherapy was initiated 3 weeks prior to study entry if the patient has recovery of blood counts and from acute toxicity of chemotherapy as described in inclusion criteria # 3.
8. Use of nitrosourea (carmustine (BCNU), lomustine (CCNU) or mitomycin - C within 6 weeks of study entry.
9. Prior surgery or Radiation Therapy (RT) within 2 weeks of study entry.
10. Patients with history of prior whole pelvic radiation will be excluded unless there is no prior history of severe thrombocytopenia (i.e. platelet nadir <10,000/mm^3)
11. Patients with history of prior high dose chemotherapy with stem cell transplant or with history of prolonged thrombocytopenia (>/= 2 weeks).
12. History of any platelet disorders including Idiopathic thrombocytopenic purpura (ITP), Thrombotic thrombocytopenic purpura (TTP) or bleeding disorders.
13. History of > 4 prior chemotherapy regimens (all platinum regimens will be counted as one regimen).
14. Patients with significant bowel dysfunction secondary to tumor (significant abdominal pain with severe constipation/diarrhea (>/= Grade 3), significant difficulty maintaining oral nutrition).
15. Patients with pre-existing neuropathy > Grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 08/04/05 to 04/09/12. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 55 participants enrolled, one participant was enrolled but was a screen failure and another three withdrew without receiving any study drug thus were excluded from the trial demographics.
Groups:
- 1 mcg/kg AMG 531 Post Chemotherapy: Cycle 1, Chemotherapy alone (Control Cycle); Beginning Cycle 2, Chemotherapy followed by 1 mcg/kg AMG 531 subcutaneously on day after chemotherapy and 2 days later (study cycle) of 21-28 day treatment cycle.
  Chemotherapy :
  1. Carboplatin [area under the concentration curve (AUC) = 11]; or
  2. Adriamycin /Ifosfamide (AI) regimens [Adriamycin (Doxorubicin) 75-90 mg/m^2 intravenous (IV), Ifosfamide 10-14 gm/m^2 IV]; or
  3. High dose Ifosfamide: 14 gm/m^2
- 10 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy: Cycle 1, Chemotherapy alone (Control Cycle); Beginning Cycle 2, Chemotherapy followed by 10 mcg/kg AMG 531 for 2 doses on Days -5 and -3 (pre doses) and on day after chemotherapy and 2 days later (post doses) of 21-28 day treatment cycle.
  Chemotherapy :
  1. Carboplatin [area under the concentration curve (AUC) = 11]; or
  2. AI regimen [Adriamycin 75-90 mg/m^2 intravenous (IV), Ifosfamide 10-14 gm/m^2 IV]; or
  3. High dose Ifosfamide: 14 gm/m^2.
Period: Overall Study
Arm/Group | 1 mcg/kg AMG 531 Post Chemotherapy | 3 mcg/kg AMG 531 Post Chemotherapy | 10 mcg/kg AMG 531 Post Chemotherapy | 10 mcg/kg Pre/Post Chemotherapy | 5 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy | 10 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy
Started | 7 | 6 | 8 | 11 | 11 | 12
Completed | 6 | 6 | 6 | 10 | 10 | 10
Not Completed | 1 | 0 | 2 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Chemotherapy Changed | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Cycle 1, Chemotherapy alone (Control Cycle); Beginning Cycle 2, Chemotherapy followed by AMG 531 subcutaneously of 21-28 day treatment cycle. There were 51 participants who received at least one dose of the study drug.
Groups:
- 1 mcg/kg AMG 531 Post Chemotherapy: Cycle 1: Chemotherapy
  Cycle 2: Chemotherapy, 1 mcg/kg AMG 531 subcutaneously on day after chemotherapy and 2 days later
- 3 mcg/kg AMG 531 Post Chemotherapy: Cycle 1: Chemotherapy
  Cycle 2: Chemotherapy, 3 mcg/kg AMG 531 subcutaneously on day after chemotherapy and 2 days later
- 10 mcg/kg AMG 531 Post Chemotherapy: Cycle 1: Chemotherapy
  Cycle 2: Chemotherapy, 10 mcg/kg AMG 531 subcutaneously on day after chemotherapy and 2 days later
- 10 mcg/kg Pre/Post Chemotherapy: Cycle 1: Chemotherapy
  Cycle 2: Chemotherapy, 10 mcg/kg AMG 531 subcutaneously on Day -5 (pre dose) and on day after chemotherapy
- 5 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy: Cycle 1: Chemotherapy
  Cycle 2: Chemotherapy, 5 mcg/kg AMG 531 for 2 doses on Days -5 and -3 (pre doses) and on day after chemotherapy and 2 days later (post doses)
- 10 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy: Cycle 1: Chemotherapy
  Cycle 2: Chemotherapy, 10 mcg/kg AMG 531 for 2 doses on Days -5 and -3 (pre doses) and on day after chemotherapy and 2 days later (post doses)
- Total: Total of all reporting groups
Arm/Group | 1 mcg/kg AMG 531 Post Chemotherapy | 3 mcg/kg AMG 531 Post Chemotherapy | 10 mcg/kg AMG 531 Post Chemotherapy | 10 mcg/kg Pre/Post Chemotherapy | 5 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy | 10 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy | Total
Number analyzed (Participants) | 6 | 6 | 6 | 11 | 10 | 12 | 51
Age, Continuous [Median (Full Range); unit: years] | 46 [27 to 60] | 50 [23 to 67] | 31 [24 to 63] | 37 [19 to 59] | 46 [33 to 61] | 49 [20 to 62] | 43 [19 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 5 | 5 | 6 | 28
  Male | 1 | 2 | 3 | 6 | 5 | 6 | 23
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 11 | 10 | 12 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events in Sequential Cohort Dose Escalation Study of AMG 531 Following Chemotherapy
Description: Number of participants experiencing an adverse event (AE) or serious adverse event (SAE) during study treatment, possible or probable related to study drug. All toxicities graded using the Common Terminology Criteria for Adverse Events version 3.0. Participation has a maximum of 6 cycles of chemotherapy on the study.
Time Frame: Toxicity assessments with each dose level/cycle (21-28 day cycle) up to 6 cycles
Population: All participants who received treatment were evaluable for toxicity; therefore 51 participants who received at least one dose of the study drug were evaluable for toxicity.
Measure: Number; unit: participants
Arm/Group | 1 mcg/kg AMG 531 Post Chemotherapy | 3 mcg/kg AMG 531 Post Chemotherapy | 10 mcg/kg AMG 531 Post Chemotherapy | 10 mcg/kg Pre/Post Chemotherapy | 5 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy | 10 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy
Number analyzed (Participants) | 6 | 6 | 6 | 11 | 10 | 12
participants
  Adverse Events, Possible or Probable | 0 | 0 | 1 | 4 | 5 | 8
  Serious Adverse Events, Possible or Probable | 0 | 0 | 1 | 0 | 2 | 0
  Total Adverse Events | 0 | 0 | 2 | 4 | 7 | 8

2. Primary Outcome: Number of Participants With Venous Thromboembolism (VTE) Related Serious Adverse Events in Sequential Cohort Dose Escalation Study of AMG 531 Following Chemotherapy
Description: Number of participants experiencing an venous thromboembolism (VTE) related serious adverse event (SAE) during study treatment, possible or probable related to study drug. All toxicities graded using the Common Terminology Criteria for Adverse Events version 3.0. Participation has a maximum of 6 cycles of chemotherapy on the study. VTE events reported are part or whole total number reported for study SAEs, not in addition to SAEs reported.
Time Frame: Toxicity assessments with each dose level/cycle (21-28 day cycle) up to 6 cycles
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1 mcg/kg AMG 531 Post Chemotherapy | 3 mcg/kg AMG 531 Post Chemotherapy | 10 mcg/kg AMG 531 Post Chemotherapy | 10 mcg/kg Pre/Post Chemotherapy | 5 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy | 10 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy
Number analyzed (Participants) | 6 | 6 | 6 | 11 | 10 | 12
participants
  Pulmonary Embolism (PE) | 0 | 0 | 1 | 0 | 1 | 0
  Deep Vein Thrombosis (DVT) | 0 | 0 | 0 | 0 | 1 | 0
  Total VTE Related SAEs | 0 | 0 | 1 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events reported once the participant received their first dose of study drug, AMG 531 in Cycle 2 up to 6 cycles. Cycles were 21 to 28 days. The total study period was from August 5, 2005 to May 11, 2012.
Arm/Group | 1 mcg/kg AMG 531 Post Chemotherapy | 3 mcg/kg AMG 531 Post Chemotherapy | 10 mcg/kg AMG 531 Post Chemotherapy | 10 mcg/kg Pre/Post Chemotherapy | 5 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy | 10 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 0/11 | 2/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 4/11 | 5/10 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mcg/kg AMG 531 Post Chemotherapy (N=6) | 3 mcg/kg AMG 531 Post Chemotherapy (N=6) | 10 mcg/kg AMG 531 Post Chemotherapy (N=6) | 10 mcg/kg Pre/Post Chemotherapy (N=11) | 5 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy (N=10) | 10 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy (N=12)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mcg/kg AMG 531 Post Chemotherapy (N=6) | 3 mcg/kg AMG 531 Post Chemotherapy (N=6) | 10 mcg/kg AMG 531 Post Chemotherapy (N=6) | 10 mcg/kg Pre/Post Chemotherapy (N=11) | 5 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy (N=10) | 10 mcg/kg AMG 531 Pre/Pre/Post/Post Chemotherapy (N=12)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flu-Like Symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin/rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pain, Bone (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) — Also includes back pain, neck pain or extremity pain
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Thrombocytosis (>/= 1,000,000/mm^3) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No